CLINICAL TRIAL: NCT07131202
Title: A Phase Ib/II, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability, Preliminary Efficacy, Pharmacokinetics, and Pharmacodynamics of FL115 in Combination With a PD-1 Monoclonal Antibody in Patients With Advanced Solid Tumors
Brief Title: A Study of FL115 in Combination With a PD-1 Antibody in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Forlong Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL115-201
Record Dates: First submitted 2025-07-21; First posted 2025-08-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined treatment (Experimental)
  Interventions: Drug: FL115+PD-1

INTERVENTIONS:
Drug: FL115+PD-1 — Combined treatment

SUMMARY:
This is an open-label, multicenter, Phase Ib/II clinical study designed to evaluate the safety, tolerability, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of FL115 in combination with the anti-PD-1 monoclonal antibody, in participants with advanced solid tumors. All enrolled participants will receive FL115 and Sintilimab via intravenous (IV) infusion. Treatment will continue until disease progression (excluding pseudoprogression), unacceptable toxicity, or other protocol-specified criteria for study or treatment discontinuation, whichever occurs first.

The study consists of two parts: a dose-escalation phase (Phase Ib) and a cohort-expansion phase (Phase II). The Phase 2 part will explore the preliminary efficacy and safety of the combination therapy in patients with advanced solid tumors across different tumor types.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older and up to 80 years old.
2. Phase 1b：Patients with specific advanced solid tumors confirmed by histology or cytology who have failed all standard therapies, have no available standard treatment options, or are currently not suitable for standard treatment.

   Phase 2：Patients with advanced solid tumors of specific types, either previously treated with or naïve to standard therapies.
3. With at least one measurable lesion (according to RECIST v1.1).
4. ECOG score: 0 - 1.
5. Expected survival period ≥ 12 weeks (judged by the investigator).
6. Sufficient organ function.
7. Voluntary written informed consent and agree to comply with all protocol-specified procedures and follow-up evaluations.
8. Fertile subjects (male and female) and their partners agree to use acceptable, investigator-approved contraception during the study-required period.

Exclusion Criteria:

If any of the following criteria are met, the subjects will be excluded from the study:

1. History of previous anti-tumor treatment:

   1. Previous use of IL-2 or IL-15 agonists, including but not limited to rhIL-15 (NCI), ALT-803 (ALTOR), NKTR-214 (Nektar).
   2. Subjects who received any anti-tumor investigational drugs, approved therapies, biologics, radiotherapy, or immunotherapy within 4 weeks before the first dose (except HRT(Hormoral Replacement Therapy), testosterone, oral contraceptives, ADT for prostate cancer, or endocrine therapy for breast cancer), endocrine therapy within 2 weeks, or palliative local radiotherapy within 14 days.
   3. Within 2 weeks before the first administration of the study drug, received traditional Chinese medicine for anti-tumor indications.
   4. Subjects who received oral fluoropyrimidines or small-molecule targeted therapies discontinued the treatment ≤2 weeks or 5 half-lives (whichever is longer) prior to the first dose of the study drug.
   5. Subjects who received mitomycin C or nitrosourea treatment discontinued the medication ≤6 weeks prior to the first dose of the study drug.
2. History of other previous treatments and toxicity recovery:

   1. Known or suspected allergies to FL115 and its excipients; known history of grade 3-4 allergic reactions to interleukin treatment or other fusion proteins.
   2. Known allergies to indomethacin, acetaminophen, diphenhydramine, ranitidine, cimetidine and/or famotidine.
   3. Received systemic immunosuppressants within 4 weeks before first dose, except for: ≤10 mg/day prednisone-equivalent, local/inhaled/nasal steroids, ≤7.5 mg/day for adrenal replacement, or one-time use for contrast allergy before imaging.
   4. Received treatment with granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), thrombopoietic agents (e.g., thrombopoietin [TPO], romiplostim, eltrombopag), or erythropoiesis-stimulating agents (e.g., erythropoietin [EPO]) within 14 days prior to screening.
   5. History of allogeneic organ or PBSC/bone marrow transplant.
   6. Received live viral vaccine within 4 weeks before first dose.
   7. Prior ≥Grade 3 or treatment-discontinuing irAEs, except for hypothyroidism, type 1 diabetes, or mild skin irAEs (excluding SJS, TEN, or severe dermatitis).
   8. All AEs from prior anti-tumor therapy have not resolved to baseline or ≤Grade 1 (per NCI CTCAE v5.0). Exceptions: hair loss (any grade) and ≤Grade 2 peripheral neuropathy are allowed; hypothyroidism that are well controlled with hormone replacement therapy or other conditions eligible per inclusion/exclusion criteria may be enrolled. Other ≤Grade 2 AEs may be allowed if deemed acceptable by the investigator and inclusion should be discussed with the sponsor's medical monitor.
3. Past medical history and surgical history:

   1. Malignant tumors of the blood system (such as acute lymphocytic leukemia, acute myeloid leukemia, myelodysplastic syndrome, chronic lymphocytic leukemia, chronic myeloid leukemia, non-Hodgkin's lymphoma, Hodgkin's lymphoma, and multiple myeloma).
   2. Subjects with active central nervous system (CNS) metastatic lesions or meningeal metastasis. Exception: Asymptomatic subjects with CNS metastatic tumors if the clinical condition is controlled.
   3. Subjects who had other malignant tumors within 2 years before screening. Subjects with curable local tumors (such as basal or squamous cell skin cancer, cervical or breast carcinoma in situ), can be included after clear cure.
   4. Have active autoimmune diseases or a history of autoimmune diseases requiring systemic steroids or immunosuppressants, such as rheumatoid arthritis, lupus, Wegener's granulomatosis, Sjogren's syndrome, IBD, multiple sclerosis, myasthenia gravis, myositis, autoimmune hepatitis, vasculitis, immune thrombocytopenia, autoimmune hemolytic anemia, or glomerulonephritis.

      Exception: subjects with well-controlled endocrine disorders treated with HRT (e.g., hypothyroidism, type 1 diabetes).
   5. Subjects had any of the following pulmonary toxic reactions/diseases in the past:

      Significantly clinically significant severe pulmonary-specific diseases, including but not limited to: pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease, history of idiopathic pulmonary fibrosis, organizing pneumonia (such as obliterative bronchiolitis), history of drug-induced pneumonia.

      Active interstitial lung disease (ILD) or interstitial pneumonia; history of requiring hormone or other immunosuppressant treatment for ILD or (non-infectious) pneumonia.

      Found by history or CT examination that there was active tuberculosis infection within 1 year before enrollment or more than 1 year ago with no regular treatment.
   6. Judged by the investigator to have uncontrollable pleural effusion, pericardial effusion, or peritoneal effusion.
   7. Have a significant clinical history of cardiovascular diseases.
   8. Underwent major surgery within 4 weeks prior to signing the informed consent form.
4. Infectious Disease History:

   1. Severe infections within 4 weeks before first dose.
   2. Any history of confirmed active HBV, HCV, HIV, or active tuberculosis infection
5. Other Conditions.

   1. Pregnant or breastfeeding women.
   2. Known, documented, or suspected substance abuse. Exceptions: Prescribed opioids for pain control or other investigator-approved, medically justified cases (pending sponsor medical lead agreement).
   3. Any other conditions deemed by the investigator to render the subject unsuitable for participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2026-12-05 (Estimated); Study Completion 2028-12-05 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerance | From screening to 30 days after last dose
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
MTD/RDE | through study completion, an average of 15 months
  Maximal Tolerance Dose/Recommended dosage expand
ORR | About 24 months
  The researchers evaluated the objective response rate (ORR) as per RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
As the research has not yet begun, we will revise the plan based on the actual situation of the research after we obtain some data.